CLINICAL TRIAL: NCT05579002
Title: Evaluation of the Functional Outcome of a Bionic Myoelectric Prosthesis (Hero Arm) in Children With Upper Limb Agenesis After One Year of Use.
Brief Title: Evaluation of the Functional Outcome of Hero Arm Prosthesis in Children After One Year of Use.
Acronym: EFPHA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hopitaux de Saint-Maurice (Other)
Responsible Party: Sponsor
Other Study IDs: CEREFAM-EFPHA-001
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Abnormality of Upper Lip
Keywords: Agenesis; Forearm; Malformation; Upper limb malformation; Prosthesis; Children; limb malformation; pediatric; Transverse agenesis of the forearm
MeSH Terms: conditions — Congenital Abnormalities; Limb Deformities, Congenital | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with unilateral upper limb malformation: Children born between 2006 and 2012, with a unilateral upper limb deformity. These children are regularly followed at CEREFAM for a unilateral upper limb deformity. During their follow-up, they were fitted with different upper limb prostheses. During a consultation with one of the CEREFAM physicians, they requested a Hero Arm prosthesis following the marketing and reimbursement in France in 2019.
  Interventions: Other: Questionnaires and tests

INTERVENTIONS:
Other: Questionnaires and tests — Application of three questionnaires:
  1. Canadian Occupational Performance Measure (CORM),
  2. a version of the Disabilities of the Arm Shoulder and Hand (DASH) modified for the child
  3. a questionnaire developed by CEREFAM
     * Two analytical and functional tests:
  1) the Action Research Arm Test (ARAT) 2) modified 400-point assessment.
  Other Names: Application of questionnaires + analytical and functional tests

SUMMARY:
The goal of this observational study is to evaluate the functional impact of using a bionic myoelectric prosthesis (Hero Arm) in children with a transverse forearm agenesis upper limb deformity, after one year of use. The Hero Arm prosthesis is the first bionic myoelectric prosthesis reimbursed in France for children.

The main objective is to Identify the functional difficulties encountered by the child related to the agenesis and which could be improved by wearing this prosthesis.

The investigators will include children born between 2006 and 2012 with a unilateral upper limb malformation. These children are regularly followed at Reference Center for Limb Malformations (CEREFAM) at the Saint-Maurice Hospitals (HSM) for a unilateral upper limb deformity. CEREFAM is currently following a large cohort of children with malformations including 143 children with transverse forearm agenesis. Of these, approximately 10% have been prescribed a Hero Arm prosthesis.

After the delivery of the Hero Arm, they are followed up in occupational therapy at HSM to learn how to use the prosthesis. This training lasts two days with an evaluation (T0). This assessment includes:

* three questionnaires: the Canadian Measure of Occupational Performance (CMOP), a version of the Disabilities of the Arm Shoulder and Hand (DASH) that has been modified to fit the child, and a questionnaire completed by the CEREFAM.
* two analytical and functional tests: the Action Research Arm Test (ARAT) and the modified 400-point assessment.

The same assessment will be performed after one year of wearing the prosthesis (T1).

This is a observational and non-interventional study. No changes have been made to the usual follow-up of the patient.

DETAILED DESCRIPTION:
Transverse forearm agenesis (TFA) is a sporadic, non-genetically based, mostly isolated congenital malformation. According to Froster-Iskenius U.G. & Baird P.A, the incidence of this condition is estimated at 1.7 per 10,000 births. This condition is characterized by a lack of partial or complete development of a limb or limb segment. In transverse forearm agenesis (TFA), the majority of the damage occurs at the proximal-middle third of the limb.

In general, with the French administration, people with TFA are not considered to be disabled. However, this malformation can have a functional impact with limitations in certain activities of daily living and in the practice of specific activities (sports, music...). Socially, some patients present a desire to be "unnoticed", especially during adolescence and early adulthood, when entering professional life, for fear of discrimination in hiring. On the other hand, some patients display their malformation and even make it their "trademark".

Currently, agenesis patients are treated by multidisciplinary teams who propose a prosthesis. The prosthesis is not indispensable, patients live with their malformation since birth and are autonomous in their daily life. There are 3 categories of prostheses: aesthetic prostheses, functional prostheses and tool prostheses.

The Hero Arm prosthesis, belonging to the functional prostheses, is the first and only bionic myoelectric prosthesis reimbursed in France for children by the Social Security since 2019. This prosthesis is designed by 3D printing by Open Bionics in England. It is a prosthesis that has a lower cost than other prostheses available on the market, which is not negligible due to the growth of the child, requiring the change of prosthesis annually. The price of a Hero Arm prosthesis is around 12,000 to 15,000 euros. This prosthesis is a departure from traditional aesthetic prosthesis models and is closer to "superhero" type prostheses. In addition, there is a variety of colors available and the appearance can be customized by the children.

Until now, no study has been done on the functional results of the Hero Arm prosthesis in à pediatric context in France.

This is the first study on the use of a new bionic myoelectric prosthesis in children in France, retrospective, allowing to evaluate the service rendered by the medical device and the impact on the quality of life of these children with congenital amputation of the forearm. This study is based on the patients of the Reference Center for Limb Malformations (CEREFAM).

Beyond the functional aspect, this study will allow to frame the prescription of this prosthesis by analyzing the service rendered for the child and their family.

ELIGIBILITY:
Inclusion Criteria:

* Children between 7 and 16 years old
* Children with a unilateral upper limb deformity
* Children with a Hero Arm bionic myoelectric prosthesis, with or without another prosthesis
* Children and parents who speak and understand French
* No objection to data collection

Exclusion Criteria:

* Children with bilateral upper limb malformation
* Children with cognitive disorders who are not able to learn to use a myoelectric prosthesis

Ages: 7 Years to 16 Years | Sex: All
Age Groups: Child
Study Population: We include children born between 2006 and 2012 with a unilateral upper limb malformation. These children are regularly followed at CEREFAM for a unilateral upper limb deformity. During their follow-up, they requested a Hero Arm prosthesis.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-01-02 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (MCRO) / change is being assessed | T0 at first use of the prosthesis and T1 at 12 months of use
  Designed to detect, from the patient's own words, the disturbances in the occupational balance that occur in the areas of personal care, productivity and leisure. This assessment highlights problems and limitations in the child's participation in meaningful activities. The child must rate his or her performance, i.e., his or her perception of his or her ability to perform the activity, as well as his or her satisfaction with this performance.
  The child can describe up to 15 problematic items with an estimation on a 10-point ordinal scale (rating) of the importance of the difficulties identified. The examiner, with the child's input, will select the 5 most important difficulties to address. The child will self-assess on a 10-point scale, for each of the selected difficulties, his/her current performance ("I am capable or not") and satisfaction ("I am happy or not"). These are meaningful activities for the child at that age.
  This measure assessed change between T0 and T1.
Disability of the Arm, Shoulder and Hand (DASH) / change is being assessed | T0 at first use of the prosthesis and T1 at 12 months of use
  It was designed to be a region-specific instrument to measure the patient's perception of symptoms and disabilities associated with any upper extremity or joint disorder. We used it as a global functional assessment of the child, to evaluate what he or she is able to do with or without a prosthesis.
  The DASH consists of 30 items that measure: (a) physical abilities (21 items); (b) symptom severity (5 items) and (c) social abilities or roles (4 items). The DASH is scored using a 5-point Likert scale that rates the individual's difficulties in the previous week.
  This measure assessed change between T0 and T1
Action Research Arm Test (ARAT) / change is being assessed | T0 at first use of the prosthesis and T1 at 12 months of use
  ARAT is a measurement scale for assessing specific changes in limb function in individuals with brain injury (the result being hemiplegia). It assesses the patient's ability to manipulate objects of various sizes, weights, and shapes and can thus be considered a measure of upper extremity-specific activity limitations.
  The ARAT is divided into four subscales: Grasping; Grasping; Pinching; and Gross Motor Skills. Each subscale is a hierarchical Guttman scale, which means that each item is given in increasing order of difficulty. In the ARAT, if the patient successfully completes the most difficult item on the subscale, this suggests that he or she will succeed on the easier items on that same subscale. Similarly, failure on any item suggests that the patient will be unable to complete the more difficult items on that subscale.
  This measure assessed change between T0 and T1

SECONDARY OUTCOMES:
The 400-point balance sheet / change is being assessed | T0 at first use of the prosthesis and T1 at 12 months of use
  This is a functional evaluation of the hand. It proposes an evaluation at 4 levels: motor skills, strength, single-handed grip, bi-manual coordination. Each test is scored out of 100.
  A modification of the 400-point assessment, involving the use of tests 3 and 4 only, was carried out at the Percy Army Training Hospital to evaluate upper limb prostheses after traumatic amputation.
  This modified version of the 400-point assessment therefore includes two parts instead of the four in the unmodified version:
  Test 3: Evaluation of single-handed grasping and moving of objects. This is a timed test, where each hand will be timed.
  Test 4: Evaluation of two-handed coordination. Non-timed test
  This measure assessed change between T0 and T1
Analytical Questionnaire / change is being assessed | T0 at first use of the prosthesis and T1 at 12 months of use
  Analytical questionnaire realized by the team of the CEREFAM of Saint Maurice.
  It is divided into 6 parts:
  1. history of the use of à prostheses and reasons for stopping using prostheses in the past
  2. assesses the child's current use of the Hero Arm prosthesis
  3. Evaluates 5 criteria for Hero Arm satisfaction (aesthetics, fluidity of movement, maintenance, use, battery)
  4. assesses 9 Hero Arm disadvantage criteria (failure, battery position discomfort, weight tolerance, dressing discomfort, pain in use, skin damage and discomfort, sweat tolerance, and noise).
  5. Evaluate how the children feel about the prosthesis with an emotion scale
  6. The sixth part includes 4 open questions
  This measure assessed change between T0 and T1

CONTACTS AND LOCATIONS:
Overall Officials: Nathaly QUINTERO-PRIGENT, Doctor, Study Director — Centre de Référence pour les Anomalies des Membres (CEREFAM)
Locations (1):
- Hôpitaux de Saint-Maurice, Saint-Maurice, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Jong IG, Reinders-Messelink HA, Janssen WG, Poelma MJ, van Wijk I, van der Sluis CK. Mixed feelings of children and adolescents with unilateral congenital below elbow deficiency: an online focus group study. PLoS One. 2012;7(6):e37099. doi: 10.1371/journal.pone.0037099. Epub 2012 Jun 8. PMID 22715362
- [Background] Kerver N, van Twillert S, Maas B, van der Sluis CK. User-relevant factors determining prosthesis choice in persons with major unilateral upper limb defects: A meta-synthesis of qualitative literature and focus group results. PLoS One. 2020 Jun 30;15(6):e0234342. doi: 10.1371/journal.pone.0234342. eCollection 2020. PMID 32603326
- [Background] Widehammar C, Pettersson I, Janeslatt G, Hermansson L. The influence of environment: Experiences of users of myoelectric arm prosthesis-a qualitative study. Prosthet Orthot Int. 2018 Feb;42(1):28-36. doi: 10.1177/0309364617704801. Epub 2017 May 4. PMID 28470129
- [Background] Cordella F, Ciancio AL, Sacchetti R, Davalli A, Cutti AG, Guglielmelli E, Zollo L. Literature Review on Needs of Upper Limb Prosthesis Users. Front Neurosci. 2016 May 12;10:209. doi: 10.3389/fnins.2016.00209. eCollection 2016. PMID 27242413
- [Result] Manero A, Smith P, Sparkman J, Dombrowski M, Courbin D, Kester A, Womack I, Chi A. Implementation of 3D Printing Technology in the Field of Prosthetics: Past, Present, and Future. Int J Environ Res Public Health. 2019 May 10;16(9):1641. doi: 10.3390/ijerph16091641. PMID 31083479